CLINICAL TRIAL: NCT03942120
Title: Post-Marketing Surveillance for Crohn's Disease Patients Treated With STELARA
Brief Title: Post-Marketing Surveillance for Crohn's Disease Participants Treated With Stelara (Ustekinumab)
Acronym: STELARA CD PMS
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108610; CNTO1275CRD4029 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants with Crohn's Disease: Participants that are diagnosed with Crohn's disease will be observed in this study who are being treated with ustekinumab under real world clinical practice. Only data available per clinical practice will be collected within this study.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Participants treated with ustekinumab under real world clinical practice will be observed in this study. No study drug will be administered as a part of this study.
  Other Names: Stelara

SUMMARY:
The purpose of post-marketing surveillance (PMS) is to assess the safety and effectiveness of ustekinumab (Stelara) for Crohn's disease participants under real world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are administered with Stelara for the first time for the indication of Crohn's disease in accordance with the label
* Participants must sign a participation agreement/informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

- Have contraindication to Stelara in accordance to the label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible participants who are being prescribed ustekinumab (Stelara) for the treatment of Crohn's disease indication will be part of this study.
Sampling Method: Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Approximately up to 3 years
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Change from Baseline in Crohn's Disease Activity Index (CDAI) Score | Baseline up to 3 years
  CDAI is a scoring system to assess the symptoms of participants with Crohn's disease (CD). It consists of 8 different CD-related factors that are summed after adjustment with a weighting factor. These 8 variables are: extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid stools, abdominal pain/cramping, and general well-being. CDAI total score ranges from 0 to 900 and a decrease over time indicates improvement in disease activity.
Change from Baseline in C-reactive Protein (CRP) Concentration | Baseline up to 3 years
  Change from baseline in CRP concentration will be assessed.
Change from Baseline in Harvey-Bradshaw Index (HBI) Score | Baseline up to 3 years
  HBI is a shorter and simpler alternative version of CDAI which consists of five parameters that allow physicians to quickly categorize the severity of Crohn's disease and detect remission. The 5 parameters are: general well-being (0-4, where higher score means lower well-being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day (score 1 per movement), abdominal mass (0=none, 1=dubious, 2=definite, 3=definite and tender), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools per day and number of complications, where higher scores indicate more severe disease and, score is presented as: less than (<)5 (remission), 5-7 (mild disease), 8-16 (moderate disease), and greater than (>)16 (severe disease).
Change from Baseline in Fecal Calprotectin Level | Baseline up to 3 years
  Change from baseline in fecal calprotectin levels will be assessed. Elevated calprotectin level in the stool indicates that inflammation is present in the intestine and the degree of elevation is associated with the severity of the inflammation.
Change from Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) | Baseline up to 3 years
  SES-CD is a simplified endoscopic scoring system to evaluate Crohn's disease activity developed as an alternative to Crohn's disease endoscopic index of severity (CDEIS). It assesses the size of mucosal ulcers, the ulcerated surface, the endoscopic extension and the presence stenosis. Each endoscopic component is scored from 0 to 3 for each segment, and a total score is derived from the sum of all the component scores (range, 0 [remission] to 60 [the most severe endoscopic activity]).
Change from Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score | Baseline up to 3 years
  SIBDQ is a simple, validated 10-item self-reported questionnaire for participants with inflammatory bowel disease to evaluate participant-reported outcomes in 4 domains- digestive symptoms (3 items), systemic symptoms (2 items), emotional disturbance (3 items), and social function (2 items). Participants rate each item on a 7-point Likert scale (1=all of the time; 2=most of the time; 3=a good bit of the time; 4=some of the time; 5=a little bit of the time; 6=hardly any of the time; 7=none of the time). Total score is calculated by adding the scores from each domain; the total score ranges from 10 to 70, where minimum score =10 (poor quality of life) and maximum score =70 (good quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (43):
- South Korea (43):
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Good Gangan Hospital, Busan
  - Pusan National University Hospital, Busan
  - Dong-A University Hospital, Busan
  - Samsung ChangWon Hospital, Changwon
  - Changwon Kyunngsang University Hospital, Changwonsi
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Dankook University Hospital, Cheonan-si
  - Hallym University Chuncehon Medical Center, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Daegu Fatima Hospital, Daegu
  - Kyongpook national university Medical center, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Koo Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Chunnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - GyeongSang National University Hospital, Jinju
  - Bucheon Soonchunhyang Hospital, Kyunggido
  - The Catholic Univ. of Korea, DaeJeon St. Mary's Hospital, Seongnam
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Pusan National University Yangsan Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Hallym University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - KyungHee University Hospital, Seoul
  - Yonsei University Severance Hospital - Dept.of Internal Medicine, Seoul
  - Gangnam Severance Hospital, Seoul
  - Ewha Woman's University Seoul Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Derived] Lee CK, Moon W, Chun J, Kim ES, Kim HW, Yoon H, Kim HS, Lee YJ, Choi CH, Jung Y, Park SC, Song GA, Lee JH, Jung ES, Kim Y, Jung SY, Choi JM, Ye BD. One-year Safety and Effectiveness of Ustekinumab in Patients With Crohn's Disease: The K-STAR Study. Inflamm Bowel Dis. 2025 May 12;31(5):1306-1316. doi: 10.1093/ibd/izae171. PMID 39096895